CLINICAL TRIAL: NCT00861445
Title: A Randomized, Double-Blind Placebo Controlled Trial to Investigate Safety and Efficacy of SPM927 in Painful Diabetic Neuropathy
Brief Title: A Trial to Investigate Safety and Efficacy of SPM927 in Painful Diabetic Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Study Director, UCB
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SP0614
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2010-07

CONDITIONS: Painful Diabetic Neuropathy
Keywords: Lacosamide, Vimpat®
MeSH Terms: conditions — Diabetic Neuropathies | interventions — 2-(acetylamino)-3-methoxy-N-(phenylmethyl)-, (2R)-; Lacosamide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: SPM927/Lacosamide
- 2 (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: SPM927/Lacosamide — SPM927 (film-coated tablets, 25/50/100mg per tablet), dosage 400mg/day, intake in the morning and in the evening, intake for 10 weeks
  Arms: 1
Other: Placebo — Placebo tablets two times a day for 10 weeks
  Other Names: SPM927; Lacosamide; Vimpat®
  Arms: 2

SUMMARY:
The primary purpose is to investigate the safety and efficacy of SPM927 in patients with Painful Diabetic Neuropathy

ELIGIBILITY:
Inclusion Criteria:

* Subject has clinically diagnosed pain attributed to diabetic distal sensory motor polyneuropathy for 1-5 years and a diagnosis of diabetes mellitus (Type I or Type II).
* Subjects must have at least moderate pain (mean pain intensity ≥ 4 out of 10 during the baseline week on Likert scale).
* subjects must have good or fair diabetic control (Hgb A1c < 10%)

Exclusion Criteria:

* Subject has other conditions that cause neuropathic pain at least as severe as the diabetic pain i.e. peripheral arterio-vascular disease.
* Subject receives treatment for seizures.
* Subject has had any amputations other than diabetically-related toe amputations.
* Subject has major skin ulcers.
* Subject has clinically significant ECG abnormalities.
* Subject is expected to take within 7 days prior to randomization and during the study: TCAs, mexiletine hydrochloride, lidoderm patch, tramadol, AEDs, dextromethorphan, opioids, capsaicin, nonsteroidal anti-inflammatory drugs, acetaminophen / paracetamol, skeletal muscle relaxants, benzodiazepines, alpha-2-agonists (e.g. clonidine), drugs indicated for sleep disturbance (e. g. zolpidem tartrate, zaleplon) and over-the-counter medications with centrally acting properties.
* Subject has laboratory values which are outside the normal range and judged by the investigator to be clinically significant.
* At study entry, subject has liver function tests values (AST, ALT,alkaline phosphatase, total bilirubin and GGT) 2 times upper limit of normal.
* subject has impaired renal function, i.e., creatinine clearance is lower than 60 mL/min.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2001-06; Primary Completion 2003-01 (Actual); Study Completion 2003-02 (Actual)

PRIMARY OUTCOMES:
The primary objective of this trial is to evaluate the efficacy of SPM 927 in reducing pain in subjects with diabetic distal sensory polyneuropathy | Assessments throughout the trial, either daily and/or at clinic visits

SECONDARY OUTCOMES:
Different qualities of neuropathic pain, sleep and activity (daily assessment during entire trial participation) | Daily assessment during entire trial participation including visits at the site
Quality of Life and the Profile of Mood States (assessment at site visits during entire trial participation) | Daily assessment during entire trial participation including visits at the site
Investigate the tolerability and safety of SPM927 (assessment during entire trial participation) | Daily assessment during entire trial participation including visits at the site
Examine the pharmacokinetics of SPM927 (assessment at all site visits during entire trial participation) | Daily assessment during entire trial participation including visits at the site

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)

REFERENCES:
- [Result] Rauck RL, Shaibani A, Biton V, Simpson J, Koch B. Lacosamide in painful diabetic peripheral neuropathy: a phase 2 double-blind placebo-controlled study. Clin J Pain. 2007 Feb;23(2):150-8. doi: 10.1097/01.ajp.0000210957.39621.b2. PMID 17237664